CLINICAL TRIAL: NCT04715854
Title: Comparison of the Addition of an Aerosol Mask Above Nasal Canula on Oxygenation in Hypoxemic Failure
Brief Title: Effect on paO2 of Adding an Aerosol Mask Above the Nasal Canulas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratory of Movement, Condorcet, Tournai, Belgium (Other)
Responsible Party: Principal Investigator, frédéric Duprez, Deputy director, clinician, laboratory of movement Condorcet Belgium, Laboratory of Movement, Condorcet, Tournai, Belgium
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: lmcondorcet
Record Dates: First submitted 2021-01-03; First posted 2021-01-20 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Hypoxemic Respiratory Failure; Emergencies; Covid19
Keywords: mask, oxygen
MeSH Terms: conditions — Respiratory Insufficiency; Emergencies; COVID-19 | interventions — Masks

STUDY DESIGN:
Intervention Model Description: One group will receive oxygen by classical nasal cannula. The second group will receive oxygen by aerosol mask associated with the nasal cannula. Afterward, the sequence will be inverted.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nasal canula (flexicare) (Active Comparator): Patients will receive oxygen by classical nasal cannula
  Interventions: Device: Mask
- Intersurgical aerosol mask with one hole closed by tape (Active Comparator): Patients will receive oxygen by classical nasal cannula associated with an aerosol mask partially closed (one lateral hole of the face mask closed by tape)
  Interventions: Device: Mask
- Intersurgical aerosol mask (Active Comparator): Patients will receive oxygen by classical nasal cannula associated with an aerosol mask
  Interventions: Device: Mask

INTERVENTIONS:
Device: Mask — addition of the mask above the nasal cannulas

SUMMARY:
This study will compare the impact of a classical aerosol mask above low-flow nasal cannula on the arterial oxygen tension in patients with COVID-19.

DETAILED DESCRIPTION:
Hospitalized patients with COVID-19 typically present with hypoxemia. In some patients, hypoxemia can be corrected with low flow nasal cannula. When placed above nasal cannula, some systems have demonstrated their interest in improving the performance of the patient's oxygen delivery. For example, two recent studies have shown that adding a Double-Trunk Mask (DTM) or Surgical Mask (SM) above nasal cannula has the potential to improve the PaO2 despite no change in oxygen output (1, 2) . However, no study has compared the effect on PaO2, of the addition of a classical aerosol mask above nasal canula.

ELIGIBILITY:
Inclusion Criteria:

Hypoxemia

Exclusion Criteria:

Hypercapnia

Confusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in PaO2 and PaCO2 | 30 minutes
  Changes in PaO2 [ Time Frame: At baseline and 30 minutes after wearing the randomized oxygen delivery system ] Oxygen tension (PaO2) in mmHg will be analyzed from a sample taken from the arterial system

SECONDARY OUTCOMES:
Respiratory frequency | 1 minute
  Change in respiratory rate [ Time Frame: At baseline, 30 minutes and 60 minutes after wearing the randomized oxygen delivery system ] Respiratory frequency is measured during one minute by visual inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Epicura, Hornu, Hainaut, Belgium